CLINICAL TRIAL: NCT06068049
Title: An Ambispective, Non-interventional, Multiple Cohort Study to Assess the Management of Osimertinib Treatment in Patients With EGFRm Non-small Cell Lung Cancer Under Real-world Conditions in Spain
Brief Title: OSIREAL - Osimertinib RWE on EGFRm NSCLC in Spain
Acronym: OSIREAL
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5162R00034
Record Dates: First submitted 2023-07-26; First posted 2023-10-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (4):
- Cohort 1: Patients diagnosed with locally advanced or metastatic NSCLC with activating EGFR mutations that received first line treatment with osimertinib (FLAURA regimen).
- Cohort 2: Patients with stage IB-IIIA NSCLC after complete tumour resection that has activating mutations in the EGFR (deletion of exon 19 or substitution of exon 21 [L858R]) that received adjuvant treatment with osimertinib (ADAURA regimen).
- Cohort 3: Patients with advanced NSCLC whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations, that received osimertinib in combination with pemetrexed and platinum-based chemotherapy for the first- line treatment (FLAURA2 regimen).
- Cohort 4: Patients with locally advanced, unresectable NSCLC treated with osimertinib, whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations and whose disease has not progressed during or following platinum-based chemoradiation therapy (LAURA regimen).

SUMMARY:
Lung cancer (LC) is the tumor responsible for the highest mortality worldwide. Lung adenocarcinoma is the major subtype of lung cancer and represents the deadliest human cancer, affecting current-, ex-, and even non-smokers.

Osimertinib is indicated as monotherapy for the first-line (1L) treatment of adult patients with locally advanced or metastatic NSCLC with activating mutations in the EGFR, for the treatment of adult patients with EGFR T790M mutation-positive locally advanced or metastatic NSCLC, for the adjuvant treatment of adult patients with NSCLC stages IB-IIIA after complete resection of the tumor that has activating mutations of the EGFR, for the treatment of adult patients with locally advanced, unresectable NSCLC whose tumours have EGFR exon 19 deletions or exon 21 substitution mutation and whose disease has not progressed during or following platinum-based chemoradiation therapy, and in combination with pemetrexed and platinum-based chemotherapy for the 1L treatment of adult patients with advanced NSCLC whose tumours have EGFR exon 19 deletions or exon 21 substitution mutations.

The FLAURA trial showed that treatment with osimertinib significantly prolongs PFS and improves overall survival (OS) compared to standard EGFR tyrosine kinase inhibitors.

The results of the ADAURA study showed a reduction in the risk of recurrence or death by 83% in stages II to IIIA, and in 80% in stages IB-IIIA. Additionally, osimertinib demonstrated a highly statistically significant improvement in DFS and HRQoL was maintained.

The FLAURA2 trial showed that 1L treatment with osimertinib-chemotherapy led to significantly longer progression-free survival than osimertinib monotherapy among patients with EGFR mutated (EGFRm) advanced NSCLC.

The LAURA trial showed that treatment with osimertinib after chemoradiotherapy resulted in significantly longer PFS than placebo among patients with unresectable stage III EGFRm NSCLC.

To date, there are no real-world data on osimertinib either in 1L treatment in locally advanced or metastatic EGFRm NSCLC nor as adjuvant treatment, in early stages of cancer, regarding effectiveness, adherence, treatment exposure and quality of life (QoL), among others, and in particular for the use of osimertinib in subpopulations less represented in pivotal trials such as elderly or patients with uncommon EGFR mutations. Furthermore, the duration of treatment in real life in Spain is also a gap, as it appears to be longer than in clinical trials, which means that there are patients who are treated beyond progression.

Therefore, this observational ambispective study based on real-world data aims to provide data on osimertinib use as adjuvant treatment in adult patients diagnosed with stages IB-IIIA EGFRm NSCLC, in 1L treatment in patients with locally advanced or metastatic EGFRm NSCLC, as consolidation treatment in patients with locally advanced, unresectable NSCLC whose tumours have EGFR exon 19 deletions or exon 21 substitution mutations and whose disease has not progressed during or following platinum-based chemoradiation therapy, and in combination with pemetrexed and platinum-based chemotherapy in patients with advanced NSCLC whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution. Specifically, the study will focus on patient characteristics, adherence, treatment exposure, administration, survival, quality of life, effectiveness and safety providing insights into osimertinib use in daily practice for patients with EGFRm NSCLC, where there are current evidence gaps.

DETAILED DESCRIPTION:
Cancer continues to be one of the leading causes of morbidity and mortality in the world. It is estimated that in the year 2020, approximately 18.1 million new cases of cancer in the world, and that this figure will increase in the next two decades to 27 million. The most frequently diagnosed tumors in the world in 2020 were those of the breast, lung (which occupies the second position), colon and rectum, prostate and stomach, all of them with more than one million cases.

Also, in Spain, cancer is one of the main causes of morbidity and mortality. It is estimated that in 2020 there were 113,054 deaths from cancer in Spain. The number of cancers diagnosed in Spain in 2022 is estimated to reach 280,100 cases according to REDECAN calculations, which represents a slight increase compared to previous years. Lung cancer (LC) is the tumor responsible for the highest mortality worldwide. After prostate cancer, it is the second most common cancer in men and, after breast cancer, in women. Lung adenocarcinoma is the major subtype of lung cancer and represents the deadliest human cancer, affecting current-, ex-, and even non-smokers.

The most frequently diagnosed cancers in Spain in 2023 will be those of the colon and rectum, breast, lung, prostate, and urinary bladder. Lung cancer is a very common cancer in Spain, however, due to its high mortality, its prevalence at five years is relatively low.

Approximately 30% of patients with non-small cell lung cancer (NSCLC) have early-stage disease that is treated with surgery. A high percentage of these patients relapse and die, so patients receive postoperative adjuvant systemic chemotherapy to increase their survival. However, the benefits of this strategy are modest. NSCLC is often associated with druggable molecular alterations that drive lung carcinogenesis. EGFR tyrosine kinase inhibitors (TKIs) have been included in treatment paradigms with the aim of improving the outcome of adjuvant therapy in patients with completely resected, EGFR mutation-positive (EGFRm+) disease.

Osimertinib is indicated as monotherapy for the first-line treatment of adult patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with activating mutations in the epidermal growth factor receptor (EGFR), for the treatment of adult patients with EGFR T790M mutation-positive locally advanced or metastatic NSCLC, for the adjuvant treatment of adult patients with NSCLC stages IB-IIIA after complete resection of the tumor that has activating mutations of the EGFR (exon 19 deletion or exon 21 substitution (L858R)), for the treatment of adult patients with locally advanced, unresectable NSCLC whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations and whose disease has not progressed during or following platinum-based chemoradiation therapy, and in combination with pemetrexed and platinum-based chemotherapy for the first-line treatment of adult patients with advanced NSCLC whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations.

The FLAURA trial showed that treatment with osimertinib significantly prolongs progression-free survival (PFS) compared to EGFR TKI comparator (median 18.9 months and 10.2 months, respectively, HR=0.46, 95% CI: 0.37, 0.57; P<0.0001) (5) and improves overall survival (OS) (HR=0.799 [95.05% CI: 0.641, 0.997]) compared to standard EGFR tyrosine kinase inhibitors (TKIs), in patients with EGFR mutation-positive advanced non-small-cell lung cancer (NSCLC). A greater proportion of patients treated with osimertinib were alive at 12, 18, 24 and 36 months (89%, 81%, 74% and 54% respectively) compared to patients treated with EGFR TKI comparator (83%, 71%, 59% and 44% respectively).

The results of the ADAURA trial showed that adjuvant treatment with osimertinib reduced the risk of recurrence or death by 83% in stages II to IIIA, and in 80% in stages IB-IIIA, compared with placebo, in patients with NSCLC with completely resected stage IB to IIIA disease and confirmed EGFR mutation. Additionally, osimertinib demonstrated a highly statistically significant improvement in disease free survival (DFS) and HRQoL was maintained. A DFS benefit favouring osimertinib over placebo was seen across all prespecified subgroups, including those based on disease stage, EGFR sensitizing mutation, ethnicity and receipt of adjuvant chemotherapy. Furthermore, the DFS benefit with osimertinib was similar in patients who had or had not received chemotherapy.

The FLAURA2 trial showed that first-line treatment with osimertinib-chemotherapy led to significantly longer progression-free survival than osimertinib monotherapy among patients with EGFR mutated advanced NSCLC . Investigator-assessed progression-free survival was significantly longer in the osimertinib-chemotherapy group than in the osimertinib group (hazard ratio for disease progression or death, 0.62; 95% confidence interval [CI], 0.49 to 0.79; P<0.001). At 24 months, 57% (95% CI, 50 to 63) of the patients in the osimertinib- chemotherapy group and 41% (95% CI, 35 to 47) of those in the osimertinib group were alive and progression-free. An objective response was observed in 83% of the patients in the osimertinib-chemotherapy group and in 76% of those in the osimertinib group; the median response duration was 24.0 months (95% CI, 20.9 to 27.8) and 15.3 months (95% CI, 12.7 to 19.4), respectively. The safety profile of osimertinib plus pemetrexed and a platinum-based agent was consistent with the established profiles of the individual agents.

The LAURA trial showed that treatment with osimertinib after chemoradiotherapy resulted in significantly longer progression-free survival than placebo among patients with unresectable stage III EGFR-mutated NSCLC. Osimertinib offered a median PFS of 39.1 months, compared with only 5.6 months with placebo (HR 0.16, 95% CI [0.10, 0.24]; P<0.0001). The percentage of patients who were alive and progression free at 12 months was 74% (95% CI, 65 to 80) with osimertinib and 22% (95% CI, 13 to 32) with placebo. The overall safety profile of osimertinib after chemoradiotherapy was consistent with the established profile of osimertinib and chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, treated with osimertinib
* Age ≥ 18 years at starts of osimertinib treatment (i.e., index date).
* Patients histologically diagnosed with EGFRm NSCLC (before index date):

  * Patients with first-line treatment with EGFRm locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy (Cohort 1).
  * Patients with stage IB-IIIA whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations, after complete tumor resection (Cohort 2).
  * Patients with advanced NSCLC whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations, that received osimertinib in combination with pemetrexed and platinum-based chemotherapy for the first-line treatment (Cohort 3).
  * Patients with locally advanced, unresectable NSCLC treated with osimertinib, whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations and whose disease has not progressed during or following platinum-based chemoradiation therapy (cohort 4).
* Provision of informed consent (for alive patients). Deceased patients who met the selection criteria when they started treatment with osimertinib could also be included in the study.

Exclusion Criteria:

* Osimertinib treatment administration in a clinical trial setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult EGFRm NSCLC patients receiving osimertinib according to SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of osimertinib in terms of median OS in patients with locally advanced or metastatic EGFRm NSCLC (Cohort 1). | From start of osimertinib treatment to death, assessed up to 6 years
  - Overall survival (OS) measured as median time from start of osimertinib treatment to death.
  The primary measure of interest is median OS and corresponding 95% confidence interval.
To evaluate the effectiveness of osimertinib in terms of 4-year rwDFS rate in patients with stages IB-IIIA EGFRm NSCLC (Cohort 2). | From start of osimertinib treatment to death, assessed up to 4 years.
  The primary measure of interest is the 4-year real world disease-free survival rate and corresponding 95% confidence interval.
  - 4-year real world disease-free survival rate for Cohort 2. (i.e., percentage of patients with clinical or radiological recurrence or death from any cause in the absence of disease recurrence 4 years after the start of osimertinib treatment, as evaluated by the treating physician according to standard clinical practice).
To evaluate the effectiveness of osimertinib in combination with pemetrexed and platinum-based chemotherapy in terms of 3-year OS in adult patients with advanced NSCLC whose tumours have EGFRm exon 19 deletions or exon 21 (L858R) substitution (Cohort 3). | From start of osimertinib treatment to death, assessed up to 3 years.
  The primary measure of interest is 3-year overall survival rate and corresponding 95% confidence interval.
  - 3-year OS rate for Cohort 3 (i.e., percentage of patients alive 3 years after the start of osimertinib treatment).
To evaluate the effectiveness of osimertinib (median rwPFS) in patients with locally advanced, unresectable NSCLC with EGFR exon 19 deletions or exon 21 (L858R) substitution mutations whose disease is stable during or after platinum-based CRT (Cohort 4). | From start of osimertinib treatment to death, assessed up to 3 years.
  - Real World Progression-free survival (rwPFS) defined as the median time from start of osimertinib treatment to clinical/radiological progression or death from any cause, in the absence of progression, as evaluated by the treating physician according to standard clinical practice.
  The primary measure of interest is median rwPFS and corresponding 95% confidence interval.

SECONDARY OUTCOMES:
To further evaluate the effectiveness of osimertinib in terms of rwPFS in patients with locally advanced or metastatic EGFRm NSCLC (Cohort 1). | From start of osimertinib to clinical/radiological progression or death from any cause, whichever came first, assesed up to 6 years
  Real World Progression-Free Survival (rwPFS) defined as the time from start of osimertinib treatment to clinical/radiological progression or death from any cause, in the basence of progression, as evaluated by the treating physician according to standard clinical practice.
  The measure of interest is the median rwPFS.
To further evaluate the effectiveness of osimertinib in terms of rwDFS rates and OS in patients with stages IB-IIIA EGFRm NSCLC (Cohort 2). | From start of osimertinib to clinical/radiological recurrence or death from any cause, whichever came first, assesed up to 4 years
  The measure of interest is the median rwDFS and rates and corresponding 95% confidence intervals.
  Overall survival (OS) measured as median time from start of osimertinib treatment to death.
  The measure of interest is the median and OS rates and corresponding 95% confidence intervals.
To further evaluate the effectiveness of osimertinib in combination with pemetrexed and platinum-based CT in terms of rwPFS and OS, in patients with advanced NSCLC whose tumours have EGFRm exon 19 deletions or exon 21 (L858R) substitution (Cohort 3). | From start of osimertinib to clinical/radiological progression or death from any cause, whichever came first, assesed up to 3 years.
  The measure of interest is the 3-year rwPFS defined as percentage of patients with clinical or radiological progression or death from any cause in the absence of disease recurrence 3 years after the start of osimertinib treatment, as evaluated by the treating physician according to standard clinical practice.
  The measure of interest are OS rates and corresponding 95% confidence intervals.
To further evaluate the effectiveness of osimertinib in terms of CNS PFS, rwTTDM and 3-year OS (Cohort 4). | From start of osimertinib to clinical/radiological progression or death from any cause, whichever came first, assessed up to 3 years.
  CNS PFS defined as the time to the earliest of CNS progression or death.
  rwTTDM defined as the time from osimertinib start date until the first date of distant metastasis or date of death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that is outside of the radiation field.
  The measures of interest are CNS PFS, rwTTDM and OS rate at 3 years and corresponding 95% confidence interval.
To describe the characteristics of osimertinib treatment administration for EGFRm NSCLC. | During osimertinib treatment, assessed up to 6 years in cohort 1 and up to 3 years in cohorts 2, 3 & 4.
  - Duration of treatment in real life, measured as time from start of osimertinib treatment to discontinuation of treatment or death from any cause in the absence of discontinuation (TTD).
  The measure of interest is discontinuation rates.
  - Real World Time to First Subsequent Therapy defined as the time from treatment initiation until the start of subsequent therapy or death (rwTFST).
  The measure of interest is discontinuation rates.
  - Frequency of dose changes and/or interruptions or reductions and their reasons.
To describe healthcare resource use (HCRU) during the osimertinib treatment for EGFRm NSCLC in real life. | During osimertinib treatment, assessed up to 6 years in cohort 1 and up to 3 years in cohorts 2, 3 & 4.
  Healthcare resources used in relation to EGFRm NSCLC and its treatment assessed by the mean number of hospitalizations (and their duration) and outpatient, pharmacy and emergency unit visits related to EGFRm NSCLC and specific tests/procedures performed.
To describe the safety profile of osimertinib in a real-world setting. | During osimertinib treatment, assessed up to 6 years in cohort 1 and up to 3 years in cohorts 2, 3 & 4
  Events of clinical interest (ECIs) (start and end date, causality, impact on treatment (i.e., requires dose reduction or interruption), adverse events that lead to osimertinib dose changes, interruptions, or permanent discontinuation, and AEs that are considered serious (including fatal events).

OTHER OUTCOMES:
To describe the effectiveness, safety and use of healthcare resources of osimertinib monotherapy in patients with locally advanced or metastatic EGFRm NSCLC (Cohort 1) who have uncommon EGFR mutations. | rwPFS from start of treatment initiation until disease progression or death; OS from treatment initiation until death from any cause.
  * rwPFS.
  * Overall survival.*
    *Overall survival (OS) measured as median time from start of osimertinib treatment to death and rates.
  * AEs that lead to osimertinib dose changes, interruptions, or permanent discontinuation, ECIs during osimertinib treatment and AEs that are considered serious (including fatal events).
  * Healthcare resources used in relation to EGFRm NSCLC and its treatment.
To describe the effectiveness, safety and use of healthcare resources of osimertinib monotherapy in elderly patients (>65 and >75 years) with locally advanced or metastatic EGFRm NSCLC (Cohorts 1, 3 & 4). | rwPFS from start of treatment initiation until disease progression or death; OS from treatment initiation until death from any cause.
  * rwPFS.
  * Overall survival.
  * AEs that lead to osimertinib dose changes, interruptions, or permanent discontinuation, ECIs during osimertinib treatment and AEs that are considered serious, including fatal events.
  * Healthcare resources used in relation to EGFRm NSCLC and its treatment.
To evaluate patient reported outcomes and experience measures (PROMs and PREMs) in EGFRm NSCLC patients treated with Osimertinib as adjuvant treatment (only applicable to cohort 2). | SATMED-Q, SF-36: at study inclusion and every 6 months. ADAQ: at study inclusion and every week during on osimertinib treatment, an average of 3 years.
  Scores on the Treatment Satisfaction with Medicines Questionnaire (SATMED-Q).
  Scores on the SF-36: 36-Item Short Form Survey. The standard version of SF-36 has a recall period of four weeks.
  Scores on the treatment adherence questionnaire (ADAQ) will be reported weekly.
  Note: these questionnaires will only be collected for patients in cohort 2 who have initiated osimertinib treatment within a maximum period of 12 months before patient inclusion in the study.
To evaluate PROMs and PREMs in patients with advanced NSCLC treated with osimertinib in combination with pemetrexed and platinum-based chemotherapy, whose tumours have EGFRm exon 19 deletions or exon 21 (L858R) substitution (Cohort 3). | SATMED-Q, SF-36: at study inclusion and every 6 months during osimertinib treatment, an average of 3 years. ADAQ: at study inclusion and every week during osimertinib treatment, an average of 3 years.
  Scores on the Treatment Satisfaction with Medicines Questionnaire (SATMED-Q).
  Scores on the SF-36: 36-Item Short Form Survey. The standard version of SF-36 has a recall period of four weeks.
  Scores on the treatment adherence questionnaire (ADAQ) will be reported weekly.
  Note: these questionnaires will only be collected for patients in cohort 3 who have initiated osimertinib treatment within a maximum period of 12 months before patient inclusion in the study.
To evaluate PROMs and PREMs in patients with locally advanced, unresectable NSCLC treated with osimertinib, with EGFR exon 19 deletions or exon 21 (L858R) mutations, whose disease is stable after platinum-based CRT (Cohort 4). | SATMED-Q, SF-36: at study inclusion and every 6 months during osimertinib treatment, an average of 3 years. ADAQ: at study inclusion and every week during osimertinib treatment, an average of 3 years.
  Scores on the Treatment Satisfaction with Medicines Questionnaire (SATMED-Q).
  Scores on the SF-36: 36-Item Short Form Survey. The standard version of SF-36 has a recall period of four weeks.
  Scores on the treatment adherence questionnaire (ADAQ) will be reported weekly.
  Note: these questionnaires will only be collected for patients in cohort 4 who have initiated osimertinib treatment within a maximum period of 12 months before patient inclusion in the study.
To describe the adherence of patients with EGFRm NSCLC treated with osimertinib under real-world conditions (Cohorts 2, 3 & 4). | ADAQ: reported at study inclusion and weekly thereafter during prospective follow-iup on osimertinib treatment, an average of 3 years.
  Adherence will be measured weekly using the Adelphi Adherence Questionnaire (ADAQ) through a mobile App managed by the company Naru Intelligence. Note: Only applicable to patients in cohorts 2, 3 and 4 who have started osimertinib treatment within a maximum period of 12 months before patient inclusion in the study.
To assess factors associated with outcomes among patients treated with osimertinib 1L (cohorts 1 & 3), and patients treated with osimertinib in the consolidation (cohort 4) or adjuvant setting (cohort 2). | rwTTD, rwTFST and CNS PFS from treatment initiation till end of treatment, start of subsequent theraypy/death or the earliest of CNS/progression, respectively. rwTTDM from date of inclusion till the first date of distant metastasis/death.
  * Overall survival.
  * rwDFS
  * rwPFS
  * rwTTD
  * rwTFST
  * rw TTDM
  * CNS PFS
  Real World Time To Discontinuation (rwTTD) defined as the time from the start of osimertinib treatment to the end of the treatment.
  Real World Time to First Subsequent Therapy (rwTFST) defined as the time from treatment initiation until the start of subsequent therapy or death.
  Real Wolrd Time to Death or Distant Metastases (rwTTDM) defined as the time from the date of inclusion until the first date of distant metastasis or date of death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that is outside of the radiation field.
  CNS PFS defined as the time to the earliest of CNS progression or death.
To describe the therapies received before and after osimertinib treatment progression or relapse. | Before and after osimertinib treatment, assesed up to 6 years in cohort 1 and up to 3 years in cohorts 2, 3 & 4.
  * Adjuvant, neoadjuvant: active drug, dose, mode of administration, duration, interruption.
  * Surgery: type, outcome (R0-R1).
  * Other treatments.
  * Therapies received after osimertinib treatment progression or relapse.

CONTACTS AND LOCATIONS:
Locations (25):
- Spain (25):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, C Rdoba
  - Research Site, Girona
  - Research Site, Gran Canaria
  - Research Site, Granada
  - Research Site, Ja N
  - Research Site, L Rida
  - Research Site, La Coru A
  - Research Site, León
  - Research Site, M Laga
  - Research Site, Madrid
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Palma
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vigo
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home